CLINICAL TRIAL: NCT01621126
Title: Neuromonitoring During the Latarjet Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jon JP Warner, Chief, MGH Shoulder Service, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011P000188
Record Dates: First submitted 2012-06-07; First posted 2012-06-18 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Shoulder Instability; Iatrogenic Nerve Injury
Keywords: Shoulder instability; Latarjet procedure; Nerve injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-op neuromonitoring (Experimental)
  Interventions: Device: Intra-operative neuromonitoring (XLTEK/NATUS EP Protektor)

INTERVENTIONS:
Device: Intra-operative neuromonitoring (XLTEK/NATUS EP Protektor) — Device: Intra-operative neuromonitoring A XLTEK/NATUS EP Protektor machine (at MGH) or a Cadwell Cascade Elite neuromonitoring machine (at BWH), both FDA approved for intra-operative neuromonitoring, will deliver the electrical stimulus applied transcranially to stimulate the motor cortex, while motor evoked responses will be recorded from different myotomes from both upper limbs. Also the same equipment will deliver electrical stimulus to stimulate peripherally the median and ulnar nerves at the wrists, with recording of the thalamocortical potentials in the scalp channels.

SUMMARY:
In a study performed by the Harvard Shoulder Service, it has been documented that there is a significant incidence of neurologic complications of the Latarjet procedure for shoulder instability. 5 out of 52 patients had neurologic complaints post-operatively. 3 of these nerve palsies were transient, however 2 had not yet recovered fully at time of latest follow-up and returned to the operating room for exploration and neurolysis of the axillary nerve and brachial plexus.

By using intra-operative neuromonitoring to determine exactly when there is a potential nerve injury during the procedure, the investigators will be able to modify what the investigators do at that step of the procedure, in order to decrease or possibly even eliminate the risk of neurologic injury.

DETAILED DESCRIPTION:
The investigators propose to study the intra-operative events which put nerves at risk during the Latarjet procedure. By using neuromonitoring to determine exactly when there is a potential nerve injury during the procedure, the investigators will be able to modify what the investigators do at that step of the procedure, in order to decrease or possibly even eliminate the risk of neurologic injury. Modifications to our surgical technique in response to events observed on neuromonitoring would include repositioning the operative shoulder and upper extremity, and repositioning or removing retractors. The investigators believe this would lead to a significant decrease in the incidence of neurologic complications post-operatively. Since this operation is usually performed on young, active patients, the benefits of reducing or eliminating these complications would have a far-reaching impact both for the individual and for society. Above all, the investigators feel that this is an important patient safety initiative.

ELIGIBILITY:
Inclusion Criteria:

* All patients of the two senior surgeons who will undergo the Latarjet procedure for shoulder instability will be considered for inclusion in the study.
* Our patients who have received prior approval from their insurance carrier to cover neuromonitoring during the surgical procedure will be enrolled.

Exclusion Criteria:

* Relative contraindications to transcranial electrical stimulation include: history of seizures, significant brain trauma, cerebral edema with mass effect, recent CVA, intracerebral devices (e.g., shunts, aneurysmal clips), skull defect and cardiac pacemaker. Patients with there conditions will be included in the study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon JP Warner, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachussetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Shah AA, Butler RB, Romanowski J, Goel D, Karadagli D, Warner JJ. Short-term complications of the Latarjet procedure. J Bone Joint Surg Am. 2012 Mar 21;94(6):495-501. doi: 10.2106/JBJS.J.01830. PMID 22318222
- [Background] Nagda SH, Rogers KJ, Sestokas AK, Getz CL, Ramsey ML, Glaser DL, Williams GR Jr. Neer Award 2005: Peripheral nerve function during shoulder arthroplasty using intraoperative nerve monitoring. J Shoulder Elbow Surg. 2007 May-Jun;16(3 Suppl):S2-8. doi: 10.1016/j.jse.2006.01.016. Epub 2006 Jul 26. PMID 17493556

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intra-op Neuromonitoring
Started | 40
Completed | 34
Not Completed | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Population: 40 subjects were enrolled; however, there were some subjects that were excluded for reasons that are explained in the published paper that resulted from this study. The total number of subjects excluded was 6, leaving 34 participants to be analyzed.
Arm/Group | Intra-op Neuromonitoring
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 30
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 28.4 [15 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Neurologic Complication Rate After Latarjet Procedure
Description: Nerve palsy of any nerve(s) in the operative upper extremity.
Time Frame: up to 24 weeks after the procedure
Measure: Number; unit: participants
Arm/Group | Intra-op Neuromonitoring
Number analyzed (Participants) | 34
participants | 7

ADVERSE EVENTS:
Arm/Group | Intra-op Neuromonitoring
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes